CLINICAL TRIAL: NCT03458299
Title: Strategies for Preventing Underage Drinking and Other Substance Use in Native American Tribal Communities
Brief Title: Strategies: Motivational Interviewing/Psychoeducation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); The Scripps Research Institute (Other)
Responsible Party: Principal Investigator, Roland Moore, Center Director and Senior Research Scientist, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AA023755 (NIH); R01AA023755 (NIH)
Record Dates: First submitted 2018-02-12; First posted 2018-03-08 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Use, Underage; Substance Use; Underage Drinking
Keywords: American Indian
MeSH Terms: conditions — Underage Drinking; Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): The MI intervention will incorporate open-ended questions, personalized feedback, and discussion about participants' alcohol use and drug, associated risk behaviors (e.g., drinking and driving), and the consequences of these behaviors. Individual MI procedures will incorporate the core principles of MI described by Miller and Rollnick, including expressing empathy, developing discrepancy, rolling with resistance, and supporting self-efficacy. Therapist interventions will be tailored to the participants' readiness to change/current stage of change (pre-contemplation, contemplation, preparation, action, maintenance, and relapse).
  Interventions: Behavioral: Motivational Interviewing
- Psychoeducation (Experimental): The Psychoeducation session will consist of therapist assisted viewing and discussion of four educational DVDs about adolescent alcohol use, drug use, and driving under the influence provided by Human Relations Media, Mount Kisco, NY (hrmvideo.com).
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Motivational Interviewing — 2 hours of motivational interviewing
  Arms: Motivational Interviewing
Behavioral: Psychoeducation — 2 hours of DVD viewing and discussion
  Arms: Psychoeducation

SUMMARY:
The goal of this research program is to implement and evaluate complementary interventions designed to address underage alcohol, marijuana, tobacco and other drug use and abuse among Native American youth residing in and around nine contiguous Indian reservations in rural portions of a Southern California county.

Component 1. Motivational Interviewing (MI) Evaluations (Identified PHI). Approximately 150 participants between 13 and 20 years of age will participate in the Motivational Interviewing (MI) intervention and one follow-up assessment over an 18 month period. Questionnaires of youth substance use and access patterns will be by phone or self-administered using paper, iPad, and web-based surveys. Formal informed consent from participants 18 and older and assent and parental/legal guardian consent will be obtained from those participants under 18.

Component 2. Psychoeducation (PE) Evaluations (Identified PHI). Approximately 150 participants between 13 and 20 years of age will participate in the Psychoeducation (PE) intervention and one follow-up assessment over an 18 month period. Questionnaires of youth substance use and access patterns will be by phone or self-administered using paper, iPad, and web-based surveys. Formal informed consent from participants 18 and older and assent and parental/legal guardian consent will be obtained from those participants under 18.

DETAILED DESCRIPTION:
Study Design. Following screening and giving informed assent/consent, eligible participants will be randomly assigned to one of two study conditions: (1) MI: Two hour session of therapist administered MI, and (2) PE: Two hour session of therapist assisted viewing and discussion of educational DVDs about adolescent alcohol use, drug use, and driving under the influence provided by Human Relations Media, Mount Kisco, NY (hrmvideo.com).

Interventions will be curriculum based in that each session will be introduced by the leader with a brief description of problems associated with underage drinking, underage binge drinking, underage tobacco and other drug use, and driving while intoxicated. Participants will be randomly assigned to the MI or PE condition, but will be able to choose an individual or group intervention format. In a preliminary study, the investigators have found that many youth prefer a group format. Both individual and group formats have been successfully used previously in this population.

Assessments will be carried out pre-intervention and once within 18 months post-intervention. Pre-intervention assessments will be carried out in person and post-intervention assessments will be done in person, by telephone, or be web-based using questionnaires developed at Brown University and previously used successfully in youth in this population. Participating youth will be paid $75 for the initial two hour intervention and $75 for completing the follow-up. The payments will be in the form of Target or other department store gift cards. All questionnaires will be available on scannable paper forms or as a web-based application to permit ease and accuracy of data transmittal to a database for evaluation.

Measures: In addition to collecting demographic data, the following measures will be used pre-intervention (MI or PE) and at follow-up: Adolescent Drinking Questionnaire (ADQ), Drug Use Questionnaire, Drinking and Drug Use Driving Scale, Tobacco Use Scale, Injury behavior checklist, Student Self Check, Relationship with Parent/Guardian - Most Important, Teen Monitoring (Chassin), Peer Substance Use, Peer Tolerance of Substance Use, Stage of Change Assessment, MI Adherence Checklist (for the MI sessions only).

Examples of potential factors include information transfer, change in beliefs, internalizing new norms, resolving ambivalence, establishing increased autonomy, empowering for change, peer modeling, and peer support. The investigators will assess 1) these change factors, 2) the participant's movement along the stages of behavior change to a new level of drinking/drug use, and 3) self-reported changes in drinking, drug use, and intoxicated driving. With these data the investigators will be able to determine not only the overall efficacy of the MI vs. PE intervention in decreasing alcohol and drug use and intoxicated driving, but also the type of behavior change (e.g., moving from pre-contemplation to action) and the variables associated with that change (e.g., internalizing new norms, increased autonomy, peer support).

The MI intervention will incorporate open-ended questions, personalized feedback, and discussion about participants' alcohol use and drug, associated risk behaviors (e.g., drinking and driving), and the consequences of these behaviors. Individual MI procedures will incorporate the core principles of MI described by Miller and Rollnick, including expressing empathy, developing discrepancy, rolling with resistance, and supporting self-efficacy. Therapist interventions will be tailored to the participants' readiness to change/current stage of change (pre-contemplation, contemplation, preparation, action, maintenance, and relapse).

In the PE intervention, participants will view all four DVDs (all DVDs available from Human Relations Media):

Session 1: Underage Drinking: Know the Facts, Know the Risks describes negative consequences of youth alcohol abuse, including deaths resulting from drunk driving, and alcohol poisoning.

Session 2: Too Much: Extreme Danger of Binge-Drinking presents information specifically about the physiology of how binge drinking can cause death, and an interview with a parent of a student who died from alcohol poisoning while partying with his friends.

Session 3: Everything You Need to Know About Substance Abuse in 22 Minutes outlines alcohol, tobacco, and other drugs' effects.

Session 4: Dying High 2: Real Stories of Drugged Driving shows consequences of driving under the influence.

Training in MI. Under the supervision of Dr. Gilder, at least six training workshops will be held with Tribal clinic study staff to deliver culturally appropriate MI to adolescent Native Americans. Workshop leaders will be Motivational Interviewing Network of Trainers (MINT) certified PhD-level trainers with expertise in working with American Indian/Alaska Native populations.

Assessment of MI fidelity. Since tribal leaders and parents, citing confidentiality and cultural concerns, stated that audio- and video-taping of MI sessions would not be acceptable, the investigators will assess the MI sessions with the Adherence Checklist - Individual and Group MI Prevention Session. The checklist contains 14 items which assess the session's process and content and the therapist's adhering to the principles of MI. Items include asking if the therapist discussed the pros and cons of changing behavior, and introduced a change plan worksheet to the participant. Therapist fidelity to MI will be assessed both during training and on an ongoing basis every 6 months during the study using the MI Adherence checklist. If the average total checklist score of adherence falls below 80%, a quality improvement program will be instituted to identify the problem(s) and correct it with additional training.

Follow-Up. The investigators believe, given the success of the preliminary pilot study in recruiting reservation youth to the initial assessment and intervention, that successful follow-up of participants represents the main potential problem for the study. These obstacles were overcome, at least in part, by 1) instituting a web-based assessment that adolescents can take any time, including free time at school; 2) keeping email and regular mail addresses of participants current; 3) increasing payment for follow-up; 4) instituting follow-up in conjunction with a program the adolescent is participating in, i.e. after school youth program, and appointments at the clinic for medical and dental services. The Tribal IRB has given permission for the web-based assessment.

This intervention study aims to recruit 150 participants to each intervention condition for a total enrollment of 300 youth participants ages 13-20 years. Evaluation will be designed to test that MI is more effective than the PE in reducing alcohol and drug use and intoxicated driving at follow-up. Evaluations to test that MI is more effective than the PE in reducing alcohol and drug use will be undertaken as follows: The primary outcome variables will be: in the previous 6 months (1) quantity x frequency of drinking, (2) frequency of binge drinking and being drunk; (3) number of days used cigarettes, other forms of tobacco, e-cigarettes and nicotine inhalant devices, cannabis, "Spice," stimulants, opiates, cough syrup, inhalants, hallucinogens, and benzodiazepines; (4) drinking or using drugs and driving and/or being a passenger in a car with a driver who has been using alcohol or drugs; (5) a negative consequences of drinking or using drugs composite score.

Descriptive statistics will be generated for each variable. Statistical analyses assessing MI vs. PE differences will be assessed as follows. For dichotomous variables, repeated-measures chi-square analyses will be used. For continuous variables, repeated measures analysis of variance (ANOVA) or analysis of covariance (ANCOVA) will be used. The Mann-Whitney Test will be used for continuous variables that are not normally distributed. Repeated measures of ordinal data for two time points will be assessed using the Wilcoxin Signed Ranks Test. With 2 groups, 150 participants in each group, an alpha = 0.01 to avoid a Type 1 error, a medium effect size for the group of dependent variables analyzed in chi-square, ANOVA, and logistic regression analyses, and a Bonferroni correction for 5 multiple comparisons in each set of analyses, the power at the projected n for chi-square, ANOVA, and logistic regression will be 0.96, 0.96, and >0.80, respectively. Power estimates were made using G*Power 3.61. If sample size permits, a larger model examining the association of selected outcome variables (e.g., frequency of bingeing and drinking/driving in the past 6 months) with independent variables (e.g., age, gender, stage of change, MI vs. PE intervention) in multiple and logistic regression models will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 13 and 20
* residing in catchment area of Tribal clinic
* ability to give informed consent/assent and absence of physical or emotional health issues sufficient to impair the ability to participate in the research

Exclusion Criteria:

* inability to give informed consent/assent or the presence of physical or emotional health issues sufficient to impair the ability to participate in the research.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
(1) Drinking QF | in the previous 6 months
  (1) quantity x frequency of drinking. [Quantity: 1, More than 10 standard drinks; 2, Between 7 and 9 standard drinks; 3, Between 5 and 6 standard drinks; 4, 4 standard drinks; 5, 3 standard drinks; 6, 2 standard drinks; 7, 1 standard drink; 8, I did not drink alcohol in the past 6 months] [Frequency: 1, Everyday; 2, 4-6 days a week, 3, 2-3 days a week; 4, once a week; 5, Less than once a week, but more than once a month, 6, Once a month 7, Less than once a month, 8, I did not drink alcohol in the past 6 months].
  Analysis: These points are inverted so that higher numbers denote higher drinking frequencies and quantities [worse outcome] and lower numbers denoted lower frequencies and quantities [better outcome]. A single quantity × frequency of drinking variable will be constructed by multiplying the frequency and quantity variables.
(2) Binge drinking/being drunk Frequency | in the previous 6 months
  (2) frequency of binge drinking and being drunk.
  Binge (female): Over the PAST 6 MONTHS, when you were drinking how many times you did drink four or more drinks (of beer, wine, or liquor)
  Binge (male): Over the PAST 6 MONTHS, when you were drinking how many times you did drink five or more drinks (of beer, wine, or liquor)
  [1. Everyday - worse outcome; 2. 4-6 days a week; 3. 2-3 days a week; 4. Once a week; 5. Less than once a week, but more than once a month; 6. Once a month; 7. Less than once a month 8. Never - better outcome].
  Drunk:
  3. Over the PAST 6 MONTHS, about how many times have you gotten drunk (drunk means you couldn't talk clearly and it was difficult to keep your balance) on alcohol?
  [1. Everyday - worse outcome; 2. 4-6 days a week; 3. 2-3 days a week; 4. Once a week; 5. Less than once a week, but more than once a month; 6. Once a month; 7. Less than once a month 8. Never - better outcome].
(3) Commercial Tobacco and Other Drug Use days | in the previous 6 months
  (3) number of days used cigarettes, other forms of tobacco, e-cigarettes and nicotine inhalant devices, cannabis, "Spice," stimulants, opiates, cough syrup, inhalants, hallucinogens, and benzodiazepines [lower numbers = better outcome, higher numbers = worse outcome]
(4) DUI/RWDD days | in the previous 6 months
  (4) drinking or using drugs and driving [During the PAST 6 MONTHS, how many times did you drive after you had been drinking? and During the PAST 6 MONTHS, how many times did you drive after you had been using drugs? - lower numbers = better outcome, higher numbers = worse outcome] and/or being a passenger in a car with a driver who has been using alcohol or drugs [During the PAST 6 MONTHS, how many times did you ride in a car with a driver who had been drinking? and 7. During the PAST 6 MONTHS, how many times did you ride in a car with a driver who had been using drugs? - lower numbers = better outcome, higher numbers = worse outcome]
(5) negative consequences of drinking or using drugs composite | in the previous 6 months
  (5) a composite score of negative consequences of drinking or using drugs.
  In the past 6 months, how many times were you injured by:
  1. Being physically attacked? (If teen response is ≥ 1, continue. If teen response is 0, skip to #2); a. How many of these times were you treated by a doctor or nurse for the injury(ies)? b. How many of these times had you been drinking alcohol about the time of the injury(ies)? c. How many of these times had you been using drugs about the time of the injury(ies)?
  2. Being in a physical fight with someone? (Do NOT include any attacks listed in previous question). a.-c. as above.
  3. Accidently getting cut? a.-c. as above.
  4. Falling? a.-c. as above.
  5. A motor vehicle accident when you were driving? a.-c. as above.
  6. A motor vehicle accident when you were not the driver? a.-c. as above. [Analysis: sum of responses; - lower numbers = better outcome, higher numbers = worse outcome]

CONTACTS AND LOCATIONS:
Overall Officials: Roland S Moore, PhD, Principal Investigator — Pacific Institute for Research and Evaluation; David A Gilder, MD, Study Director — The Scripps Research Institute
Locations (1):
- Southern California Tribal Health Center, Valley Center, California, United States

IPD SHARING:
Plan to Share IPD: No
Without explicit IRB approval, it is the policy of the IRBs overseeing this project to not share data which is personally identifiable or could reasonably lead to deductive disclosure of the identities of individual subjects. Without explicit IRB approval, it is the policy of the Southern California Tribal Health Center, The Scripps Research Institute, and the Prevention Research Center to not share data, whether personally identifiable or not, which could cause significant social, political, or legal harm to research subjects or the communities from which they come.